CLINICAL TRIAL: NCT03900598
Title: A Phase 1, First-in-Human, Open-Label Study of the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-67856633, an Inhibitor of MALT1, in Participants With NHL and CLL
Brief Title: A Study of JNJ-67856633 in Participants With Non-Hodgkin's Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108587; 67856633LYM1001 (Other: Janssen Research & Development, LLC); 2018-003549-40 (EudraCT Number); 2024-512734-15-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Dose Escalation): JNJ-67856633 (Experimental): Participants will receive JNJ-67856633 until disease progression, intolerable toxicity, withdrawal of consent, or the investigator or sponsor decision. Subsequent dose levels will be assigned by the sponsor using an adaptive dose escalation strategy based on all available safety, pharmacokinetic (PK), and biomarker data.
  Interventions: Drug: JNJ-67856633
- Part 2 (Cohort Expansion): JNJ-67856633 (Experimental): Participants will receive JNJ-67856633 at the recommended Phase 2 dose (RP2D) determined in Part 1.
  Interventions: Drug: JNJ-67856633

INTERVENTIONS:
Drug: JNJ-67856633 — JNJ-67856633 capsule will be administered orally.

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose regimen or the maximum tolerated dose of JNJ-67856633 in participants with relapsed/ refractory B-cell non-Hodgkin lymphoma and chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
Non-Hodgkin lymphoma (NHL) represents a diverse set of diseases. Among them diffuse large B-cell lymphoma (DLBCL) represents the most common subtype of NHL, accounting for 30 percent (%) to 40% of all newly diagnosed cases. Mucosa-associated lymphoid tissue lymphoma translocation protein 1 (MALT1) is a key mediator of the nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kappaB) signaling pathway and has been shown to play a critical role in different types of lymphoma, including activated B cell-like (ABC) subtype of diffuse large B-cell lymphoma (DLBCL). JNJ-67856633 is a MALT1 inhibitor and will be administered orally. The study will evaluate the following: Dose Escalation (Part 1): One or more recommended Phase 2 dose (RP2Ds) of JNJ-67856633. Cohort Expansion (Part 2): JNJ-67856633 is well tolerated and achieves antitumor responses at the RP2D. The study consists of screening phase (less than or equal to 28 days before first dose), treatment phase (from Cycle 1 Day 1 till end of treatment visit [within 30 (+7) days after the last dose]) and post-treatment phase. A prescreening period may also apply to participants in select cohorts in Part 2. The total study duration will be approximately 4 years and 11 months. Efficacy assessments will include radiographic image assessments, positron emission tomography scan, bone marrow assessment, endoscopy or colonoscopy etc. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Cardiac parameters within the following range: corrected QT interval (QTc intervals corrected using Fridericia's formula [QTcF]) less than or equal to (<=)480 milliseconds based on the average of triplicate assessments performed no more than 5 minutes apart (plus minus [+-]3 minutes)
* Women of childbearing potential must have a negative highly sensitive serum (Beta human chorionic gonadotropin) at screening and prior to the first dose of study drug, and until 30 days after the last dose
* In addition to the user-independent, highly effective method of contraception, a male or female condom with or without spermicide is required, example, condom with spermicidal foam/gel/film/cream/suppository. Male condom and female condom should not be used together (due to risk of failure with friction)
* Men must wear a condom when engaging in any activity that allows for passage of ejaculate to another person. Male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak

Exclusion Criteria:

* Known active central nervous system (CNS) involvement for dose escalation and specific expansion cohorts as determined by the study evaluation team (SET)
* Prior solid-organ transplantation
* Either of the following: a) Received an autologous stem cell transplant less than or equal to (<=)3 months before the first dose of study drug. b) Prior treatment with allogenic stem cell transplant <=6 months before the first dose of study drug, has evidence of graft versus host disease, or requires immunosuppressant therapy for graft versus host disease within the last 4 weeks
* History of malignancy (other than the disease under study in the cohort to which the participant is assigned) within 1 year prior to the first administration of study drug. Exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy which in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 1 year before the first dose of study drug. Concomitant malignancies that are unlikely to progress and/or preclude evaluation of study endpoints may be allowed after discussion with the Study Responsible Physician
* Prior treatment with a mucosa-associated lymphoid tissue lymphoma translocation protein 1 (MALT1) inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Part 1: Dose-Limiting Toxicity (DLT) | Approximately 21 days
  The DLTs are based on drug related adverse events and defined as any of the following events: any toxicity that would require discontinuation of treatment; and/or hematological / non-hematological toxicity of Grade 3 or higher.
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 4 years and 11 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

SECONDARY OUTCOMES:
JNJ-67856633 Plasma Concentrations | Up to 4 years and 11 months
  Concentration assessment will be done to evaluate the effect of JNJ-67856633.
Part 1 and Part 2: Overall Response Rate (ORR) | Up to 4 years and 11 months
  ORR is defined as the percentage of participants who have a partial response (PR) and complete response (CR) according to the International Workshop on Chronic Lymphocytic Leukemia (iwCLL), non-Hodgkin lymphoma and Waldenstrom macroglobulinemia response criteria.
Part 1 and Part 2: Complete Response Rate | Up to 4 years and 11 months
  Complete response rate is defined as the percentage of participants who achieve a best response of CR according to the iwCLL, non-Hodgkin lymphoma and Waldenstrom macroglobulinemia response criteria.
Part 1 and Part 2: Time to Response (TTR) | Up to 4 years and 11 months
  TTR is defined for participants who achieved PR or CR as the time from the first dose of study drug to first response of PR or CR.
Part 1 and Part 2: Duration of Response (DoR) | Up to 4 years and 11 months
  DoR is defined for participants who achieved PR or CR as the time between the date of initial documentation of PR or CR to the date of first documented evidence of disease progression or death, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (47):
- United States (6):
  - City of Hope, Duarte, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson, Houston, Texas
- Australia (4):
  - Monash Medical Centre, Clayton
  - Peter MacCallum Cancer Centre, Melbourne
  - Linear Clinical Research Ltd, Nedlands
  - Scientia Clinical Research, Randwick
- China (4):
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Institute of Hematology & Blood Disease Hospital Chinese Academy of Medical Science, Tianjin
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- France (8):
  - Hopital Claude Huriez, Lille
  - CHU de Nantes hotel Dieu, Nantes
  - Groupe Hospitalier Pitie Salpetriere, Paris
  - Institut Curie, Paris
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - CHU Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitatsklinikum Munster, Münster
  - Universitatsklinikum Ulm, Ulm
- Alexandra General Hospital of Athens, Athens, Greece
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Azienda Opedaliero-Universitaria Policlinico Sant'orsola Malpighi di Bologna, Bologna
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
- Japan (5):
  - National Cancer Center Hospital, Chūōku
  - Tokai University Hospital, Isehara
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Okayama University Hospital, Okayama
  - The Cancer Institute Hospital of JFCR, Tokyo
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hospital de Vall D'Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency